CLINICAL TRIAL: NCT02149940
Title: Feasibility of Pharmaceutical Interventions in Elderly Heart Failure Patients: a Pilot Study.
Brief Title: Feasibility of Pharmaceutical Interventions in Elderly Heart Failure Patients.
Acronym: RASP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S55301
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
Keywords: Elderly; Frailty; Polypharmacy; Medication review; Clinical pharmacy services
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clinical pharmacy intervention (Experimental)
  Interventions: Other: heart-failure related pharmaceutical intervention

INTERVENTIONS:
Other: heart-failure related pharmaceutical intervention

SUMMARY:
Heart failure therapies (e.g. beta blockers) have been successful in decreasing mortality rates, as well as diminishing hospitalizations. Also, pharmacist collaboration has been shown to have a beneficial impact on heart failure related outcomes. Regardless, a high residual event rate is to be noted.

In our pilot study, we wished to document whether a clinical pharmacist could still play a role in the heart failure management of an elderly inpatient heart failure population.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* diagnosis of previous or new heart failure based on signs and symptoms as defined by the 'European Society of Cardiology guidelines on acute and chronic heart failure'
* diagnosis had to be confirmed by a recent echocardiogram

Exclusion Criteria:

* not Dutch speaking
* treatment restrictions had been applied on admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
the number of heart-failure related pharmaceutical interventions | during hospital stay (average of 14 days)

SECONDARY OUTCOMES:
acceptance rate of the pharmaceutical interventions | during hospital stay (average of 14 days)
clinical feasibility of the accepted interventions | during hospital stay (average of 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Karolien Walgraeve, PharmD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lorenz R Van der Linden, PharmD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Jos Tournoy, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Flemish Brabant, Belgium

REFERENCES:
- [Derived] Walgraeve K, Van der Linden L, Flamaing J, Fagard K, Spriet I, Tournoy J. Feasibility of optimizing pharmacotherapy in heart failure patients admitted to an acute geriatric ward: role of the clinical pharmacist. Eur Geriatr Med. 2018 Feb;9(1):103-111. doi: 10.1007/s41999-017-0019-x. Epub 2018 Jan 4. PMID 34654283